CLINICAL TRIAL: NCT07144423
Title: Neuroendoscopy-assisted Drainage Versus Burr Hole Drainage for Chronic Subdural Hematoma: A Multicenter Randomized Controlled Trial, URANUS
Brief Title: Neuroendoscopy-assisted Drainage Versus Burr Hole Drainage for Chronic Subdural Hematoma
Acronym: URANUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2025027
Record Dates: First submitted 2025-07-29; First posted 2025-08-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; Neuroendoscopy-assisted Drainage; Burr Hole Drainage; Recurrence Rate; Neurological Outcome
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The design is open labeled with only the investigators for postoperative follow-up evaluation, the outcome assessors, and data analysts being blinded in all 24 centers. Before outcome assessment begins at every follow-up evaluation, the patients will be reminded not to reveal any information about their group allocation. If details of group allocation can be detected by the investigator during follow-ups, another blinded researcher will replace to evaluate outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroendoscope-assisted hematoma drainage (Experimental): Under the guidance of a visualized neuroendoscope, the hematoma is thoroughly irrigated and evacuated.
  Interventions: Procedure: Endoscope-assisted hematoma drainage
- Burr hole hematoma drainage (Other): The hematoma cavity is irrigated intraoperatively until the drainage fluid becomes clear.
  Interventions: Procedure: Burr hole hematoma drainage

INTERVENTIONS:
Procedure: Endoscope-assisted hematoma drainage — The procedure of endoscope-assisted hematoma drainage is performed under local anesthesia with sedation or general anesthesia. During the operation, a single burr hole is drilled at the midpoint of the thickest layer of the hematoma cavity as shown on CT scan. A bone flap measuring 2.0 cm × 2.0 cm is then created using a milling cutter. Under the guidance of a visualized neuroendoscope, the hematoma is thoroughly irrigated and evacuated. A subdural drainage tube is inserted, and postoperatively, continuous subdural drainage of the hematoma is maintained until the drainage ceases naturally or the drainage tube is removed at a maximum of 48 hours postoperatively to terminate the drainage.
  Arms: Neuroendoscope-assisted hematoma drainage
Procedure: Burr hole hematoma drainage — The procedure of burr hole drainage is performed under local anesthesia with sedation or general anesthesia. During the operation, a single burr hole is drilled at the midpoint of the thickest layer of the hematoma cavity as indicated by CT scan. A subdural drainage tube is then inserted. The hematoma cavity is irrigated intraoperatively until the drainage fluid becomes clear. Postoperatively, continuous subdural drainage of the hematoma is maintained until the drainage ceases naturally or the drainage tube is removed at a maximum of 48 hours postoperatively to terminate the drainage.
  Arms: Burr hole hematoma drainage

SUMMARY:
Chronic subdural hematoma (CSDH) is a frequent condition in neurosurgery, leading to fluid accumulation between the meninges, brain compression, neurological dysfunction, and potentially herniation. The efficacy of treatments and their long-term outcomes remain uncertain, with no established standard. Notably, neuroendoscopy-assisted hematoma evacuation, in contrast to burr-hole drainage, enables direct visualization and thorough removal of the hematoma, thereby minimizing residue, lowering recurrence rates, and shortening drainage duration. This study will undertake a multicenter trial to compare these two methods and determine the superior treatment approach for CSDH.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is a common disease in neurosurgery. It is generally considered to be a closed fluid collection situated between the dura mater and arachnoid mater, formed by blood or blood degradation products. This collection causes a local mass effect, compressing adjacent brain tissue and leading to varying degrees of neurological dysfunction. In severe cases, it can induce brain herniation, endangering the patient's life. In recent years, despite the availability of various pharmacological and surgical treatment options for CSDH, the efficacy and long-term prognosis of these treatment methods and strategies remain not entirely clear, and a standardized treatment approach has yet to be established. Neuroendoscopy-assisted hematoma drainage is one of the treatment methods for CSDH, but its current application is not widespread. The core of this method involves neurosurgeons directly observing the hematoma structure during surgery with the assistance of a neuroendoscope, enabling them to thoroughly irrigate and aspirate the hematoma under direct vision and sever hematoma septations. This approach enhances the hematoma clearance rate, ultimately reducing the amount of postoperative hematoma residue. Compared with conventional burr-hole drainage, neuroendoscopy-assisted burr-hole drainage reduces the recurrence rate of CSDH and shortens the duration of postoperative drainage. This study aims to conduct a multicenter randomized controlled trial comparing neuroendoscopy-assisted hematoma drainage with burr-hole drainage, with the objective of scientifically and rigorously determining the optimal clinical treatment strategy for CSDH.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (18 years to 90 years) presenting with clinical symptoms and neurological deficits of CSDH.
2. CSDH verified on cranial computed tomography or magnetic resonance imaging.
3. Written informed consent from patients or their next of kin according to the patient's cognitive status.

Exclusion Criteria:

1. No clinical symptoms correlating with chronic subdural hematoma.
2. Lack of mass effect and midline shift < 5 mm on the radiological image, or no need surgery judged clinically by neurosurgeons.
3. Previous surgery for CSDH during the past 6 months.
4. Previous intracranial surgery for any other neurological disorder.
5. Poor medication conditions or the presence of severe comorbidities so that surgery cannot be tolerated, or follow-up cannot be completed.
6. Severe coagulopathy or a high risk of life-threatening bleeding (including any one of the following three criteria: prothrombin time or activated partial thromboplastin time prolonged by more than 10 seconds; international normalized ratio > 3.0; absolute platelet count < 100×109/L).
7. Postoperative compliance is suspected to be insufficient for 3-month follow-up visit.
8. Reproductive-age women without verified negative pregnancy testing.
9. Participating in another research.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate within 3 months after operation | From operation up to 3 months postoperatively
  To compare the difference in recurrence rate at 3 months postoperatively between the two groups.

SECONDARY OUTCOMES:
Mortality rate within 3 months after operation | From operation up to 3 months postoperatively
  To compare the difference in mortality rate at 3 months postoperatively between the two groups.
Change of Modified Rankin Scale (MRS) between groups from baseline to 3 months after operation | "Day 0", "Day 2", "Month 1", "Month3" after operation
  Modified Rankin Scale ranges from score 1 to 6, and higher scores mean a worse clinical outcome, where score 1 indicates normal daily functionality and score 6 indicates death.
Change of Markwalder Grading Scale (MGS) between groups from baseline to 3 months after operation | "Day 0", "Day 2", "Month 1", "Month3" after operation
  Markwalder Grading Scale ranges from grade 0 to 4, and higher scores mean a worse neurological outcome, where grade 0 indicates normal neurological function and grade 4 indicates coma.
Change of Quality of life assessment (EQ-5D-5L) between groups from baseline to 3 months after operation | "Day 0", "Day 2", "Month 1", "Month3" after operation
  A standardized instrument, EuroQoL 5-Dimension 5-Level (EQ-5D-5L) questionnaire, will be used as a generic measure of health related quality of life. The questionnaire contains 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension rates across five levels, including 'No problems-Slight problems-Moderate problems-Severe problems-Unable to'postoperatively between the two groups.
Rate of complications and adverse events between groups within 3 months | From operation up to 3 months postoperatively
  Rate of complications and adverse events between the two groups within 3 months.
Postoperative drainage time | immediately after the procedure
  To compare the difference in length of postoperative drainage between the two groups.
Length of hospitalization | immediately after the procedure
  To compare the difference in length of hospitalization between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Guoyi Gao, MD, Principal Investigator — Beijing Tiantan Hospital; Liang Wu, MD, Study Director — Beijing Tiantan Hospital
Locations (24):
- China (24):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Shantou central hosital, Shantou, Guangdong
  - People's Hospital of Longhua, Shenzhen, Shenzhen, Guangdong
  - Liuzhou worker's Hospital, Liuchow, Guangxi
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Nanning First People's Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi University of Traditional Chinese Medicine, Nanning, Guangxi
  - Wuzhou Gongren Hospital, Wuzhou, Guangxi
  - Hebei University of Engineering Affiliated Hospital, Handan, Hebei
  - Xingtai Central Hospital, Xingtai, Hebei
  - Changde First People's Hospital, Changde, Hunan
  - People's Hospital of Xiangxi Prefecture, Hunan Province, Jishou, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Heji Hospital affiliated with Changzhi Medical College, Changzhi, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Shanxi Provincial People's Hospital,Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - Mianyang 404 Hospital, Mianyang, Sichuan
  - the First People'S Hospital of Yibin, Yibin, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Pu'er People's Hospital, Pu'er, Yunnan
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
This study plans to share de-identified individual participant data (IPD) six months after the publication of its core findings, aiming to enhance transparency and foster scientific collaboration in the field. The shared data will encompass: ① clinical indicators at baseline and follow-up (e.g., demographic characteristics, laboratory tests, outcome events); ② records of experimental interventions (grouping, surgical protocols); and ③ exclusion of identifiable information (names, precise birth dates, addresses, etc.). The data will be stored in an encrypted institutional data repository (or a public repository such as Figshare), and access will be granted only after the signing of a Data Use Agreement (DUA).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing will be opened 6 months after the completion of the study, with a duration of 5 years.
Access Criteria: Access to IPD is available to collaborators within the original research consortium. External researchers may apply via a formal request to the principal investigator (PI), including a rationale for access, proposed analysis plan, and confirmation of compliance with institutional review board (IRB) requirements. All users must sign a data usage agreement prior to receiving data.

REFERENCES:
- [Background] Abouzari M, Rashidi A, Rezaii J, Esfandiari K, Asadollahi M, Aleali H, Abdollahzadeh M. The role of postoperative patient posture in the recurrence of traumatic chronic subdural hematoma after burr-hole surgery. Neurosurgery. 2007 Oct;61(4):794-7; discussion 797. doi: 10.1227/01.NEU.0000298908.94129.67. PMID 17986941
- [Background] Asghar M, Adhiyaman V, Greenway MW, Bhowmick BK, Bates A. Chronic subdural haematoma in the elderly--a North Wales experience. J R Soc Med. 2002 Jun;95(6):290-2. doi: 10.1258/jrsm.95.6.290. PMID 12042376
- [Background] Bakheet MF, Pearce LA, Hart RG. Effect of addition of clopidogrel to aspirin on subdural hematoma: meta-analysis of randomized clinical trials. Int J Stroke. 2015 Jun;10(4):501-5. doi: 10.1111/ijs.12419. Epub 2014 Dec 3. PMID 25472690
- [Background] Banks JL, Marotta CA. Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke. 2007 Mar;38(3):1091-6. doi: 10.1161/01.STR.0000258355.23810.c6. Epub 2007 Feb 1. PMID 17272767
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Mar 17:1-8. doi: 10.3171/2016.8.JNS16134.test. Online ahead of print. PMID 28306417
- [Background] Frati A, Salvati M, Mainiero F, Ippoliti F, Rocchi G, Raco A, Caroli E, Cantore G, Delfini R. Inflammation markers and risk factors for recurrence in 35 patients with a posttraumatic chronic subdural hematoma: a prospective study. J Neurosurg. 2004 Jan;100(1):24-32. doi: 10.3171/jns.2004.100.1.0024. PMID 14743908
- [Background] Jablawi F, Kweider H, Nikoubashman O, Clusmann H, Schubert GA. Twist Drill Procedure for Chronic Subdural Hematoma Evacuation: An Analysis of Predictors for Treatment Success. World Neurosurg. 2017 Apr;100:480-486. doi: 10.1016/j.wneu.2017.01.037. Epub 2017 Jan 19. PMID 28109862
- [Background] Kudo H, Kuwamura K, Izawa I, Sawa H, Tamaki N. Chronic subdural hematoma in elderly people: present status on Awaji Island and epidemiological prospect. Neurol Med Chir (Tokyo). 1992 Apr;32(4):207-9. doi: 10.2176/nmc.32.207. PMID 1378564
- [Background] Kurabe S, Ozawa T, Watanabe T, Aiba T. Efficacy and safety of postoperative early mobilization for chronic subdural hematoma in elderly patients. Acta Neurochir (Wien). 2010 Jul;152(7):1171-4. doi: 10.1007/s00701-010-0627-4. Epub 2010 Mar 25. PMID 20336332
- [Background] Leroy HA, Aboukais R, Reyns N, Bourgeois P, Labreuche J, Duhamel A, Lejeune JP. Predictors of functional outcomes and recurrence of chronic subdural hematomas. J Clin Neurosci. 2015 Dec;22(12):1895-900. doi: 10.1016/j.jocn.2015.03.064. Epub 2015 Aug 8. PMID 26260114
- [Background] Liu W, Bakker NA, Groen RJ. Chronic subdural hematoma: a systematic review and meta-analysis of surgical procedures. J Neurosurg. 2014 Sep;121(3):665-73. doi: 10.3171/2014.5.JNS132715. Epub 2014 Jul 4. PMID 24995782
- [Background] Lu J, Shen D, Hu F, Zhou J, Lan F, Guo D, Liu T. An improved electronic twist-drill craniostomy procedure with post-operative urokinase instillation in treating chronic subdural hematoma. Clin Neurol Neurosurg. 2015 Sep;136:61-5. doi: 10.1016/j.clineuro.2015.05.037. Epub 2015 Jun 3. PMID 26067723
- [Background] Miles LA, Greengard JS, Griffin JH. A comparison of the abilities of plasma kallikrein, beta-Factor XIIa, Factor XIa and urokinase to activate plasminogen. Thromb Res. 1983 Feb 15;29(4):407-17. doi: 10.1016/0049-3848(83)90244-x. PMID 6344314
- [Background] Mori K, Maeda M. Surgical treatment of chronic subdural hematoma in 500 consecutive cases: clinical characteristics, surgical outcome, complications, and recurrence rate. Neurol Med Chir (Tokyo). 2001 Aug;41(8):371-81. doi: 10.2176/nmc.41.371. PMID 11561347
- [Background] Nakaguchi H, Tanishima T, Yoshimasu N. Factors in the natural history of chronic subdural hematomas that influence their postoperative recurrence. J Neurosurg. 2001 Aug;95(2):256-62. doi: 10.3171/jns.2001.95.2.0256. PMID 11780895
- [Background] Neils DM, Singanallur PS, Wang H, Tracy P, Klopfenstein J, Dinh D, Elwood PW, Fassett D, McCall T, Lin J, Tsung A. Recurrence-free chronic subdural hematomas: a retrospective analysis of the instillation of tissue plasminogen activator in addition to twist drill or burr hole drainage in the treatment of chronic subdural hematomas. World Neurosurg. 2012 Jul;78(1-2):145-9. doi: 10.1016/j.wneu.2011.08.032. Epub 2011 Nov 7. PMID 22120294
- [Background] Qiu S, Zhuo W, Sun C, Su Z, Yan A, Shen L. Effects of atorvastatin on chronic subdural hematoma: A systematic review. Medicine (Baltimore). 2017 Jun;96(26):e7290. doi: 10.1097/MD.0000000000007290. PMID 28658127
- [Background] Robinson RG. Chronic subdural hematoma: surgical management in 133 patients. J Neurosurg. 1984 Aug;61(2):263-8. doi: 10.3171/jns.1984.61.2.0263. PMID 6737050
- [Background] Santarius T, Hutchinson PJ. Chronic subdural haematoma: time to rationalize treatment? Br J Neurosurg. 2004 Aug;18(4):328-32. doi: 10.1080/02688690400004845. PMID 15702829
- [Background] Santarius T, Kirkpatrick PJ, Ganesan D, Chia HL, Jalloh I, Smielewski P, Richards HK, Marcus H, Parker RA, Price SJ, Kirollos RW, Pickard JD, Hutchinson PJ. Use of drains versus no drains after burr-hole evacuation of chronic subdural haematoma: a randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1067-73. doi: 10.1016/S0140-6736(09)61115-6. PMID 19782872
- [Background] Shapey J, Glancz LJ, Brennan PM. Chronic Subdural Haematoma in the Elderly: Is It Time for a New Paradigm in Management? Curr Geriatr Rep. 2016;5:71-77. doi: 10.1007/s13670-016-0166-9. Epub 2016 Mar 23. PMID 27213133
- [Background] Stanisic M, Pripp AH. A Reliable Grading System for Prediction of Chronic Subdural Hematoma Recurrence Requiring Reoperation After Initial Burr-Hole Surgery. Neurosurgery. 2017 Nov 1;81(5):752-760. doi: 10.1093/neuros/nyx090. PMID 28379528
- [Background] Weigel R, Schmiedek P, Krauss JK. Outcome of contemporary surgery for chronic subdural haematoma: evidence based review. J Neurol Neurosurg Psychiatry. 2003 Jul;74(7):937-43. doi: 10.1136/jnnp.74.7.937. PMID 12810784
- [Background] Yu GJ, Han CZ, Zhang M, Zhuang HT, Jiang YG. Prolonged drainage reduces the recurrence of chronic subdural hematoma. Br J Neurosurg. 2009 Dec;23(6):606-11. doi: 10.3109/02688690903386983. PMID 19922274
- [Background] Zhang Y, Chen S, Xiao Y, Tang W. Effects of Dexamethasone in the Treatment of Recurrent Chronic Subdural Hematoma. World Neurosurg. 2017 Sep;105:115-121. doi: 10.1016/j.wneu.2017.05.135. Epub 2017 May 31. PMID 28578110